CLINICAL TRIAL: NCT02659462
Title: Cardio Pulmonary Exercise Testing in Patients Post the Fontan Palliation in Comparison With Patients With Repaired Congenital Heart Disease and Healthy Volunteers.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0124-15-RMB CTIL
Record Dates: First submitted 2015-11-22; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Fontan Palliation; Congenital Heart Disease
Keywords: Repaired Congenital Heart Disease; Cardio Pulmonary Exercise Testing; Fontan; Fontan Palliation; functional capacity
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients post Fontan palliation for single ventricular hear: Cardio Pulmonary Exercise Testing
  Interventions: Other: Cardio Pulmonary Exercise Testing
- Subjects post surgical correction of congenital heart disease: Cardio Pulmonary Exercise Testing
  Interventions: Other: Cardio Pulmonary Exercise Testing
- Healthy patients: Cardio Pulmonary Exercise Testing
  Interventions: Other: Cardio Pulmonary Exercise Testing

INTERVENTIONS:
Other: Cardio Pulmonary Exercise Testing — Cardio Pulmonary Exercise Testing

SUMMARY:
prospective cardio respiratory evaluation for patients post the Fontan palliation for single ventricle, compared to subjects post successful cardiac repaired surgery compared to healthy volunteers in order to evaluate the functional capacity and the primary etiology for reduction in functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Children at age of 8-25 post fontan palliation
* Patients With Repaired Congenital Heart Disease without chronic lung disease
* Healthy patients ate age of 8-25

Exclusion Criteria:

* Patients with chronic lung disease
* Pregnant women
* Patients with acute active disease or chronic disease that may affect the exercise function

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. 15 patients post the Fontal palliation for single ventricular heart
  2. 15 subjects post surgical correction of congenital heart disease.
  3. 15 healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Comparing Cardio Pulmonary Exercise function between the three groups in the study | one year

CONTACTS AND LOCATIONS:
Locations (1):
- RAMBAM health care center, Haifa, Israel

REFERENCES:
- [Background] Rhodes J, Ubeda Tikkanen A, Jenkins KJ. Exercise testing and training in children with congenital heart disease. Circulation. 2010 Nov 9;122(19):1957-67. doi: 10.1161/CIRCULATIONAHA.110.958025. No abstract available. PMID 21060085
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257